CLINICAL TRIAL: NCT05020041
Title: Change Physical Activity and School Play Space. Randomized Study Protocol.
Acronym: Play&Cognition
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Universidad Autónoma de Chile (Other)
Collaborators: Ministry of Sport, Chile (Unknown)
Responsible Party: Principal Investigator, Natalia Bustamante, Principal Investigator, PhD Natalia Bustamante-Ara, Universidad Autónoma de Chile
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 01-20
Record Dates: First submitted 2021-05-05; First posted 2021-08-25 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Cognitive Function; Physical Activity; Children; Behavior, Child
MeSH Terms: conditions — Motor Activity; Child Behavior | interventions — Exercise; Neuropsychological Tests

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The implementation of painted games will consist of adapting a space destined for recreation, designing a psychomotor circuit that does not require contact between peers, or manipulation of objects to maintain COVID-19 sanitary and safety protocols.
  The schools in the intervention group will receive the online educational talk aimed at schoolchildren and a talk aimed at Physical Education teachers.
  Interventions: Behavioral: Physical activity
- Control (No Intervention): The schools participating in the control group will receive an online educational talk aimed at promoting healthy habits and the benefits of physical activity inside and outside the school environment.

INTERVENTIONS:
Behavioral: Physical activity — The schools in the intervention group will receive the online educational talk aimed at schoolchildren and a talk aimed at Physical Education teachers, given that they are fundamental for the development of habits in the school stage; besides, painted games will be implemented in the school playground.
  The implementation of painted games will consist of adapting a space destined for recreation, designing a psychomotor circuit that does not require contact between peers or manipulation of objects in order to maintain COVID-19 sanitary and safety protocols. The psychomotor circuit includes a line circuit, a jumping sequence game, and a letter spiral. All the games will be implemented in a space within the educational establishment to which the students will have access during recess. The game designs involve activities to develop motor patterns such as jumping with different supports, running, and dynamic balance.
  Other Names: Cognitive function
  Arms: Intervention

SUMMARY:
Physical activity is a factor that contributes to a motor and cognitive development in early childhood. Currently, childhood obesity has grown steadily in Chile. This study aims to evaluate the impact of a school environmental intervention on the physical activity and cognitive functions in 1st-grade schoolchildren during the COVID-19 pandemic. The study will use a randomized experimental design with a sample of 300 schoolchildren divided into a control and an intervention group (n=150 each group). Sociodemographic characteristics and lifestyle of the schoolchildren will be obtained through a questionnaire answered by parents/guardians. Cognitive function will be evaluated using the TENI test by tablet and physical activity will be measured during 7 consecutive days using accelerometers (Actigraph GT3X and wGT3X-BT). Both groups will receive a lecture aimed at schoolchildren. Teachers of the intervention group will also receive a talk regarding the intervention that will take place in their school environment, which includes a circuit of psychomotor games painted on the recess playground floor. ANCOVA analysis will be performed, adjusted for age and sex; then, a multivariate linear regression model will be applied considering the significant variables and adjustment. The significance level will be p<.05. SPSSv25 and R version 3.14 will be used for the analyses. The intervention is expected to contribute to the increase of physical activity favoring the school environment within a context of vulnerability and with a low-cost initiative

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria for the participating students are a) children enrolled in 1st-grade in municipal schools in the city of Talca; b) without impediments to physical activity; c) able to understand an order considering their age; d) residents in the commune of Talca; and e) with a commitment not to change school or residence during the duration of the project.

Exclusion Criteria:

* The exclusion criteria are presenting any medical condition that prevents the development of the evaluations and/or presenting any behavioral disorder condition.

Ages: 5 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 300 (Estimated)
Dates: Start 2021-07-22 (Actual); Primary Completion 2021-09 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Physical activity | change baseline up to 5 months
  Accelerometry data will be valid if they present ≥ 3 days of measurement with a minimum of 9 hours of use per day.
Cognitive function | change baseline up to 5 months
  The battery is composed of 8 games to assess the functioning of attention, visuospatial and visuomotor development, memory system, language, and executive functions in children aged 3 to 9 years. Test, TENI.

SECONDARY OUTCOMES:
Flowmetry | change baseline up to 5 months
  Flowmetry will be analyzed using the mean of three measurements recorded with the pediatric Mini wright (400l/m).
Hand grip strength | change baseline up to 5 months
  Manual grip strength will be assessed three times on the dominant arm using a digital dynamometer (TKK504) fitted to the palm of the schoolchild's hand

CONTACTS AND LOCATIONS:
Overall Officials: Natalia Bustamante-Ara, PhD, Principal Investigator — Universidad Autónoma de Chile
Locations (1):
- Universidad Autónoma de Chile, Talca, Maule Region, Chile

IPD SHARING:
Plan to Share IPD: No